CLINICAL TRIAL: NCT01035346
Title: Evaluation Of The Antipyretic Efficacy Of Ibuprofen Sodium Tablets In Subjects With An Uncomplicated Acute Infection
Brief Title: Study Evaluating The Efficacy Of A Novel Ibuprofen Formulation On Fever In Patients With An Uncomplicated Acute Infection
Status: Terminated | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: AH-09-12
Record Dates: First submitted 2009-12-08; First posted 2009-12-18 (Estimated); Results first posted 2012-08-21 (Estimated); Last update posted 2012-08-21 (Estimated); Status verified 2012-07

CONDITIONS: Infection
Keywords: Fever; antipyretic; uncomplicated acute viral infection; uncomplicated acute bacterial infections
MeSH Terms: conditions — Infections; Fever | interventions — Ibuprofen

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- A (Experimental)
  Interventions: Drug: Ibuprofen
- B (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Ibuprofen — Single dose of a novel ibuprofen formulation (equal to 400mg ibuprofen)
  Arms: A
Drug: Placebo — Single dose of a placebo
  Arms: B

SUMMARY:
This single-dose trial will evaluate the efficacy of a novel ibuprofen formulation compared to placebo in patients with a fever due to an uncomplicated acute infection.

ELIGIBILITY:
Inclusion Criteria:

* Subjects diagnosed with a fever secondary to an uncomplicated acute viral or bacterial infection.
* Oral temperature measurement from 100 to 104 degrees Fahrenheit.
* Onset of fever 3 days or less.
* Otherwise good health.

Exclusion Criteria:

* Fever secondary to a chronic underlying medical condition or serious infection.
* Currently taking antibiotics or antivirals.
* Currently taking any medication which may interfere with the assessment of fever.
* Pregnancy or breast-feeding.
* Any serious medical or psychiatric disorder.

Ages: 12 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2010-01; Primary Completion 2011-05 (Actual); Study Completion 2011-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Pfizer CT.gov Call Center, Study Director — Pfizer
Locations (5):
- United States (5):
  - Pfizer Investigational Site, Cypress, California
  - Pfizer Investigational Site, Westlake Village, California
  - Pfizer Investigational Site, Omaha, Nebraska
  - Pfizer Investigational Site, Pittsburgh, Pennsylvania
  - Pfizer Investigational Site, Salt Lake City, Utah

REFERENCES:
- [Derived] Jayawardena S, Leyva R, Kellstein D. Safety of a novel formulation of ibuprofen sodium compared with standard ibuprofen and placebo. Postgrad Med. 2015 Jan;127(1):33-7. doi: 10.1080/00325481.2015.993268. Epub 2014 Dec 15. PMID 25526232
- See also: To obtain contact information for a study center near you, click here. — https://trialinfoemail.pfizer.com/pages/landing.aspx?StudyID=AH-09-12&StudyName=Study%20Evaluating%20The%20Efficacy%20Of%20A%20Novel%20Ibuprofen%20Formulation%20On%20Fever%20In%20Patients%20With%20An%20Uncomplicated%20Acute%20Infection

RESULTS

PARTICIPANT FLOW:
Groups:
- Placebo: Single oral dose of 2 placebo tablets matched to ibuprofen sodium 256 milligram (mg) tablet.
- Ibuprofen Sodium: Single oral dose of 2 ibuprofen sodium 256 mg tablets, equivalent to 400 mg ibuprofen.
Period: Overall Study
Arm/Group | Placebo | Ibuprofen Sodium
Started | 7 | 9
Completed | 7 | 9
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Placebo: Single oral dose of 2 placebo tablets matched to ibuprofen sodium 256 mg tablet.
- Total: Total of all reporting groups
Arm/Group | Placebo | Ibuprofen Sodium | Total
Number analyzed (Participants) | 7 | 9 | 16
Age Continuous [Mean (Standard Deviation); unit: years] | 31.4 (15.3) | 37.3 (17.9) | 34.8 (16.5)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 4 | 6
  Male | 5 | 5 | 10
Body Temperature [Mean (Standard Deviation); unit: Degrees Fahrenheit] | 100.99 (0.83) | 100.58 (0.66) | 100.76 (0.74)

OUTCOME MEASURES:

1. Primary Outcome: Time-weighted Sum of The Temperature Differences From Baseline Through Hour 6 (STEMPD 0-6)
Description: STEMPD 0-6 was defined as time-weighted sum of temperature differences over 6 hours, weighted by the time elapsed between each 2 consecutive time points. Temperature difference was defined as baseline temperature minus post-baseline temperature at each time point, where positive value indicated improvement in body temperature.
Time Frame: 0 to 6 hours
Population: Intent-to-treat (ITT) population included all randomized participants who received study medication and provided a baseline temperature assessment.
Measure: Mean (Standard Deviation); unit: Degrees Fahrenheit
Arm/Group | Placebo | Ibuprofen Sodium
Number analyzed (Participants) | 7 | 9
Degrees Fahrenheit | 3.0 (6.3) | 10.8 (4.9)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; Treatment difference (Ibuprofen sodium-Placebo) and corresponding 95 percent (%) confidence interval (CI) were calculated based on Least-squares (LS) means from the Analysis of Variance (ANOVA) model; Test type: Superiority or Other; p = 0.228, ANOVA — p-value was calculated using ANOVA model with treatment and baseline temperature terms. Statistical testing was done at 5% significance level (2-sided); Least-squares (LS) mean difference = 8.33, 95% CI 2-sided [-7.94 to 24.60]

2. Secondary Outcome: Time-weighted Sum of The Temperature Differences From Baseline Through Hour 4 and Hour 8 (STEMPD 0-4 and STEMPD 0-8)
Description: STEMPD 0-4 and STEMPD 0-8 were defined as the time-weighted sum of temperature differences over 4 hours and 8 hours, weighted by the time elapsed between each 2 consecutive time points. Temperature difference was defined as baseline temperature minus post-baseline temperature at each time point, where positive value indicated improvement in body temperature.
Time Frame: 0 to 4, 0 to 8 hours
Population: ITT population included all randomized participants who received study medication and provided a baseline temperature assessment.
Measure: Mean (Standard Deviation); unit: Degrees Fahrenheit
Arm/Group | Placebo | Ibuprofen Sodium
Number analyzed (Participants) | 7 | 9
Degrees Fahrenheit
  STEMPD 0-4 | 1.7 (3.9) | 6.7 (2.9)
  STEMPD 0-8 | 5.7 (9.4) | 13.4 (7.3)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; STEMPD 0-4: Treatment difference (Ibuprofen sodium-Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.171, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 5.99, 95% CI 2-sided [-3.99 to 15.97]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen Sodium; STEMPD 0-8: Treatment difference (Ibuprofen sodium-Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.354, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 8.96, 95% CI 2-sided [-14.78 to 32.69]

3. Secondary Outcome: Change From Baseline in Temperature at Hours 0.25, 0.5, 1, 2, 4, 6 and 8
Description: Change from baseline in temperature was calculated as baseline temperature minus post-baseline temperature at each time point, where positive value indicated improvement in body temperature.
Time Frame: Baseline, 0.25, 0.5, 1, 2, 4, 6, 8 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Degrees Fahrenheit
Arm/Group | Placebo | Ibuprofen Sodium
Number analyzed (Participants) | 7 | 9
Degrees Fahrenheit
  0.25 hours | 0.4 (0.4) | 0.4 (0.3)
  0.5 hours | 0.5 (0.4) | 0.7 (0.4)
  1 hour | 0.3 (0.7) | 1.2 (0.7)
  2 hours | 0.8 (1.0) | 1.9 (0.9)
  4 hours | 0.3 (1.5) | 2.0 (0.9)
  6 hours | 0.7 (1.5) | 2.1 (1.3)
  8 hours | 1.3 (1.7) | 1.3 (1.9)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; 0.25 hours: Treatment difference (Ibuprofen sodium-Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.576, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = -0.15, 95% CI 2-sided [-0.84 to 0.54]
Statistical Analysis 2: Comparison: Placebo vs Ibuprofen Sodium; 0.5 hours: Treatment difference (Ibuprofen sodium-Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.502, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 0.18, 95% CI 2-sided [-0.50 to 0.87]
Statistical Analysis 3: Comparison: Placebo vs Ibuprofen Sodium; 1 hour: Treatment difference (Ibuprofen sodium-Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.116, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 1.31, 95% CI 2-sided [-0.51 to 3.12]
Statistical Analysis 4: Comparison: Placebo vs Ibuprofen Sodium; 2 hours: Treatment difference (Ibuprofen sodium-Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.161, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 1.58, 95% CI 2-sided [-0.98 to 4.14]
Statistical Analysis 5: Comparison: Placebo vs Ibuprofen Sodium; 4 hours: Treatment difference (Ibuprofen sodium-Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.215, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 1.87, 95% CI 2-sided [-1.66 to 5.41]
Statistical Analysis 6: Comparison: Placebo vs Ibuprofen Sodium; 6 hours: Treatment difference (Ibuprofen sodium-Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.388, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 1.17, 95% CI 2-sided [-2.18 to 4.52]
Statistical Analysis 7: Comparison: Placebo vs Ibuprofen Sodium; 8 hours: Treatment difference (Ibuprofen sodium-Placebo) and corresponding 95% CI were calculated based on LS means from the ANOVA model; Test type: Superiority or Other; p = 0.849, ANOVA — [p-value comment as in outcome 1, analysis 1]; LS mean difference = 0.31, 95% CI 2-sided [-3.98 to 4.61]

4. Secondary Outcome: Time to Treatment Failure
Description: Median time of dropping out of the participants from the study due to lack of efficacy or use of rescue medication, whichever comes first.
Time Frame: 0 to 8 hours
Population: as for outcome 2
Measure: Median (95% Confidence Interval); unit: hours
Arm/Group | Placebo | Ibuprofen Sodium
Number analyzed (Participants) | 7 | 9
hours | NA [NA to NA] — Data was not summarized, as median time to treatment failure for placebo group was greater than 8 hours (study duration) therefore 95% CI was not estimable. | NA [NA to NA] — Data was not summarized, as median time to treatment failure for ibuprofen sodium group was greater than 8 hours (study duration) therefore 95% CI was not estimable.

5. Secondary Outcome: Cumulative Percentage of Participants With Treatment Failure
Description: Percentage of participants who withdrew from the study due to lack of efficacy or received rescue medication.
Time Frame: 0.25, 0.5, 1, 2, 4, 6, 8 hours
Population: as for outcome 2
Measure: Number; unit: percentage of participants
Arm/Group | Placebo | Ibuprofen Sodium
Number analyzed (Participants) | 7 | 9
percentage of participants
  0.25 hours | 0.0 | 0.0
  0.5 hours | 0.0 | 0.0
  1 hour | 0.0 | 0.0
  2 hours | 0.0 | 0.0
  4 hours | 0.0 | 0.0
  6 hours | 0.0 | 0.0
  8 hours | 0.0 | 11.1
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; 8 hours: Treatment difference (Ibuprofen sodium-Placebo) and its associated CI were calculated based on Cochran-Mantel-Haenszel (CMH) adjusted proportion and the corresponding standard errors; Test type: Superiority or Other; p = 0.378, Cochran-Mantel-Haenszel — p-value was calculated using CMH general association test using table scores. Statistical testing was done at 5% significance level (2-sided); difference in proportion = 11.11, 95% CI 2-sided [-10.67 to 32.89]

6. Secondary Outcome: Global Assessment of Study Medication as an Antipyretic
Description: Global assessment of study medication was performed at the 8-hours time point or immediately before taking rescue medication (if necessary). It was scored on a 5-point categorical scale where 0=poor, 1=fair, 2=good, 3=very good, and 4=excellent.
Time Frame: 8 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen Sodium
Number analyzed (Participants) | 7 | 9
units on a scale | 1.8 (1.5) | 2.5 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; Treatment difference (Ibuprofen sodium-Placebo) and the associated CI were calculated based on the weighted Gamma statistic; Test type: Superiority or Other; p = 0.324, Cochran-Mantel-Haenszel — p-value was calculated using CMH test with modified ridit scores. Statistical testing was done at 5% significance level (2-sided); Mean Difference (Final Values) = 0.48, 95% CI 2-sided [-0.30 to 1.27]

7. Secondary Outcome: Rating of Study Medication Relative to Usual Medication
Description: Rating of study medication was performed at the 8-hours time point or immediately before taking rescue medication (if necessary). It was scored on a 5-point categorical scale where 0=poor, 1=fair, 2=good, 3=very good, and 4=excellent.
Time Frame: 8 hours
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Ibuprofen Sodium
Number analyzed (Participants) | 7 | 9
units on a scale | 1.5 (1.4) | 2.4 (1.1)
Statistical Analysis 1: Comparison: Placebo vs Ibuprofen Sodium; [analysis description as in outcome 6, analysis 1]; Test type: Superiority or Other; p = 0.210, Cochran-Mantel-Haenszel — [p-value comment as in outcome 6, analysis 1]; Mean Difference (Final Values) = 0.53, 95% CI 2-sided [-0.12 to 1.18]

ADVERSE EVENTS:
Arm/Group | Placebo | Ibuprofen Sodium
Serious Adverse Events (participants affected / at risk) | 0/7 | 0/9
Other Adverse Events (participants affected / at risk) | 1/7 | 3/9
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (N=7) | Ibuprofen Sodium (N=9)
Cold sweat (General disorders) | 0 | 1
Fatigue (General disorders) | 0 | 1
Malaise (General disorders) | 0 | 1
Pain (General disorders) | 1 | 0
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 1 | 0
Pruritus (Skin and subcutaneous tissue disorders) | 0 | 1

LIMITATIONS AND CAVEATS:
Definitive conclusion could not be made due to early termination of study, due to low enrollment rate, and small number of enrolled participants.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Pfizer has the right to review disclosures, requesting a delay of less than 60 days. Investigator will postpone single center publications until after disclosure of pooled data (all sites), less than 12 months from study completion/termination at all participating sites. Investigator may not disclose previously undisclosed confidential information other than study results.